CLINICAL TRIAL: NCT00419510
Title: Genetic Counseling for Breast Cancer Susceptibility in African American Women
Brief Title: Genetic Counseling in African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 704355; DAMD17-00-1-0262
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Genetic counseling; BRCA1 and BRCA2; African American
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1

INTERVENTIONS:
Behavioral: Culturally Tailored Genetic Counseling

SUMMARY:
The objectives of this study are to develop a Culturally Tailored Genetic (CTGC) protocol for African American women and evaluate its impact on decision making and satisfaction about BRCA1/2 testing, quality of life, and cancer control practices compared to Standard Genetic Counseling (SGC). A secondary objective of this study is to identify African American women who are most and least likely to benefit from CTGC vs. SGC.

DETAILED DESCRIPTION:
Five to 10% of all breast cancer cases have been attributed to two breast ovarian cancer susceptibility genes called BRCA1 and BRCA2 (BRCA1/2). Genetic counseling and testing for BRCA1/2 mutations is now available through clinical research programs using standard counseling protocols. The goal of pre test counseling is to facilitate informed decision making about whether to be tested and to prepare participants for possible outcomes. The goal of post test counseling is to provide information about risk status, recommendations for surveillance, and options for prevention. However, previous research suggests that African American and Caucasian women differ in their attitudes about and responses to pre test education and counseling. Increasingly, cultural beliefs and values are being recognized as important factors in genetic counseling. Despite recommendations to increase the cultural sensitivity of breast cancer risk counseling, such programs have not been developed or evaluated. Therefore, the purpose of this study is to develop a Culturally Tailored Genetic Counseling (CTGC) protocol for African American women and evaluate its impact on psychological functioning and health behaviors compared with Standard Genetic Counseling (SGC) in a randomized clinical trial.

1. To evaluate the relative impact of CTGC vs. SGC on decision making and satisfaction about BRCA1/2 testing. Compared to SGC, CTGC will lead to higher rates of test acceptance and satisfaction with testing decisions. These effects will be mediated by increases in perceived benefits and decreases in perceived limitations and risks of genetic testing.
2. To evaluate the impact of CTGC vs. SGC on quality of life and health behaviors following BRCA1/2 testing. Compared to SGC, CTGC will lead to larger decreases in general and cancer specific distress, greater increases in adherence to cancer screening guidelines, and lower rates of prophylactic surgery. Reductions in psychological distress will be mediated by increased use of spiritual coping strategies.

Secondary Aim

To identify African American women who are most and least likely to benefit from CTGC vs. SGC. We predict that the relative benefits of CTGC will be greatest for women with greater endorsement of African American cultural values and those identified as BRCA1/2 carriers.

ELIGIBILITY:
Inclusion Criteria:

* Female
* African American or Black
* 5% to 10% prior probability of having a BRCA1 or BRCA2 mutation

Exclusion Criteria:

* Men
* Individuals who are not African American or Black

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2003-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Psychological functioning
Cancer screening behaviors
Cancer risk reduction behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Chanita Hughes-Halbert, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Halbert CH, Kessler L, Collier A, Weathers B, Stopfer J, Domchek S, McDonald JA. Low rates of African American participation in genetic counseling and testing for BRCA1/2 mutations: racial disparities or just a difference? J Genet Couns. 2012 Oct;21(5):676-83. doi: 10.1007/s10897-012-9485-y. Epub 2012 Jul 12. PMID 22790832
- [Derived] Halbert CH, Kessler L, Troxel AB, Stopfer JE, Domchek S. Effect of genetic counseling and testing for BRCA1 and BRCA2 mutations in African American women: a randomized trial. Public Health Genomics. 2010;13(7-8):440-8. doi: 10.1159/000293990. Epub 2010 Mar 17. PMID 20234119